CLINICAL TRIAL: NCT04752540
Title: A Phase I, Single-dose, Parallel Group Study to Assess the Pharmacokinetics of Olorofim in Subjects With Hepatic Impairment
Brief Title: A Phase I Study to Assess the Pharmacokinetics of Olorofim in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F901318-01-16
Record Dates: First submitted 2021-02-11; First posted 2021-02-12 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild hepatic impairment (Experimental): 120 mg olorofim
  Interventions: Drug: Olorofim
- Moderate hepatic impairment (Experimental): 60 to 120 mg olorofim
  Interventions: Drug: Olorofim
- Normal hepatic function (Active Comparator): 120 mg olorofim
  Interventions: Drug: Olorofim

INTERVENTIONS:
Drug: Olorofim — single oral dose
  Other Names: F901318

SUMMARY:
A single oral dose study to investigate the PK and safety of olorofim in mild and moderately hepatically impaired subjects compared to subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 70 years of age inclusive, at the time of signing the informed consent.
* Body weight ≥50 kg and BMI within the range 18 to 35 kg/m2 (inclusive
* Subjects with mild hepatic impairment will have grade A Child-Pugh score of 5 to 6 at screening and Day -1:
* Subjects with moderate hepatic impairment: will have grade B Child-Pugh score of 7 to 9 at screening and Day -1
* Subjects with normal liver function must be in good health, as determined by a medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations
* Subjects with normal liver function are matched by gender, age (±10 years) and BMI (± 20%) to at least one hepatically impaired subject.

Exclusion Criteria:

* Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risk of participating in the study
* Subjects with any history of convulsion (other than childhood febrile convulsion before the age of 6 years).
* Subjects who have any clinically significant allergic disease (excluding mild or seasonal allergies such as contact dermatitis or hay fever) as determined by the Investigator.
* Subjects with a history of or any concomitant active malignancy.
* Subjects with a history of drug or alcohol abuse.
* Subjects with, or with a history of, any clinically significant neurological, renal, cardiovascular, psychiatric, respiratory, metabolic, endocrine, ocular (including minor trauma), hematological, or other major disorders as determined by the Investigator.
* Subjects with signs or symptoms consistent with a COVID-19 infection at screening or Day -1
* Hepatically impaired subjects with liver transplantation, autoimmune liver disease, or drug-induced liver damage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2021-10-24 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to the time of the last quantifiable concentration (AUC 0-t) | 0-96 hours
Maximum Observed Plasma Concentration (Cmax) | 0-96 hours

SECONDARY OUTCOMES:
Time to Reach Maximum Plasma Concentration (Tmax) | 0-96 hours
Apparent Elimination Half Life (t1/2) | 0-96 hours
Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC 0-inf) | 0-96 hours
Number of Participants With Treatment-Emergent Adverse Events | 10 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orange County Research Centre, Tustin, California
  - Orlando Clinical Research Centre, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No